CLINICAL TRIAL: NCT00317980
Title: Phase IV Randomized Controlled Clinical Trial to Evaluate the Safety and Efficacy of Low-Dose Pentavalent Antimony Compared to the Standard Dose in Patients With Cutaneous Leishmaniasis Caused by Leishmania (Viannia)Braziliensis
Brief Title: Safety and Efficacy of Low-Dose Pentavalent Antimony for Treatment of Cutaneous Leishmaniasis
Acronym: Lowdosesb
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Gustavo S Romero MD, Nucleo de Medicina Tropical, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMT-LD-CP-2006
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous leishmaniasis; Leishmania braziliensis; Pentavalent antimony; Meglumine antimoniate
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose (Experimental): Meglumine antimoniate 5 mg/kg/d for 20 days
  Interventions: Drug: Meglumine antimoniate
- Standard dose (Active Comparator): Meglumine antimoniate 15 mg/kg/d for 20 days
  Interventions: Drug: Meglumine antimoniate

INTERVENTIONS:
Drug: Meglumine antimoniate — Meglumine antimoniate 5mg/kg/d for 20 days
  Other Names: Glucantime
  Arms: Low dose
Drug: Meglumine antimoniate — Meglumine antimoniate 15 mg/kg/d for 20 days
  Other Names: Glucantime
  Arms: Standard dose

SUMMARY:
The purpose of this study is to determine whether low-dose pentavalent antimony is equally effective when compared to the standard-dose regimen in patients with cutaneous leishmaniasis. The study will be done in a field clinic in the state of Bahia, Brazil.

DETAILED DESCRIPTION:
The first-choice drug for the treatment of cutaneous leishmaniasis in Brazil is the pentavalent antimonial meglumine antimoniate. The treatment with meglumine antimoniate is toxic and at least some of the more relevant adverse events associated with that drug are dose-dependent. Recently, some research developed in Brazil has shown evidence that lower doses of pentavalent antimony are equally efficacious as compared to the standard-dose regimen. That evidence has been obtained in patients from the State of Rio de Janeiro who were infected by Leishmania (Viannia) braziliensis. The purpose of the study is to evaluate the safety and efficacy of the low-dose pentavalent antimony regimen in patients with cutaneous leishmaniasis infected by Leishmania (Viannia) braziliensis living in a rural area of the State of Bahia, Brazil, where cutaneous leishmaniasis is highly endemic. The usefulness of the study is based on the possibility to reduce the toxicity observed during treatment and the treatment costs.

The main comparison of the therapeutic response is going to be made between two groups composed of an equal number of properly randomized patients with localized cutaneous leishmaniasis treated with any of the following drug schemes:

* Meglumine antimoniate (calculated dose based on the concentration of pentavalent antimony) 5 mg/kg/d intravenous for 20 days
* Meglumine antimoniate (calculated dose based on the concentration of pentavalent antimony) 15 mg/kg/d intravenous for 20 days

The clinical outcomes of cure or failure will be evaluated until the third month of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Presence of 1 to 9 cutaneous lesions clinically compatible with leishmaniasis
* Disease duration of 2 to 20 weeks
* Positive leishmanin skin test
* Parasitological diagnosis confirmed through culture or genus-specific polymerase chain reaction (PCR) for Leishmania spp

Exclusion Criteria:

* History of past episode of leishmaniasis
* Mucosal disease
* Disseminated disease
* Use of drugs with anti-leishmanial activity
* Contraindications for using pentavalent antimony:

  * pregnancy
  * renal failure
  * heart failure
  * hepatic failure
* Other diseases:

  * active tuberculosis
  * hanseniasis

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Actual)
Dates: Start 2006-02; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Proportion of clinically cured patients at the third month after treatment | Three months after treatment
Proportion of patients with epithelialized lesions | Three months after treatment

SECONDARY OUTCOMES:
Proportion of patients with adherence to the protocol prescribed drug | 30 days
Proportion of patients with adverse events | 30 days after treatment
Proportion of patients with late failure after the first three months of follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo S Romero, MD, Principal Investigator — University of Brasilia
Locations (1):
- Núcleo de Medicina Tropical, University of Brasilia, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Oliveira-Neto MP, Schubach A, Mattos M, Goncalves-Costa SC, Pirmez C. Treatment of American cutaneous leishmaniasis: a comparison between low dosage (5 mg/kg/day) and high dosage (20 mg/kg/day) antimony regimens. Pathol Biol (Paris). 1997 Jun;45(6):496-9. PMID 9309267
- [Background] Oliveira-Neto MP, Schubach A, Mattos M, Goncalves-Costa SC, Pirmez C. A low-dose antimony treatment in 159 patients with American cutaneous leishmaniasis: extensive follow-up studies (up to 10 years). Am J Trop Med Hyg. 1997 Dec;57(6):651-5. doi: 10.4269/ajtmh.1997.57.651. PMID 9430521